CLINICAL TRIAL: NCT00812617
Title: Effects of Mineral Water Consumption on Serum Lipid Parameters: a Double-Blind, Randomized Controlled Trial
Brief Title: Effects of Mineral Water Consumption on Serum Lipid Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: Hita Tenryosui Co., Ltd. (Unknown)
Responsible Party: Fumiko higashikawa, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: eki-77
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
MeSH Terms: interventions — Mineral Waters

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Mineral water 1 (Experimental)
  Interventions: Dietary Supplement: Mineral water (Hita, Oita, Japan)
- Mineral water 2 (Experimental)
  Interventions: Dietary Supplement: Mineral water (Aso-gun, Kumamoto, Japan)

INTERVENTIONS:
Dietary Supplement: Mineral water (Hita, Oita, Japan)
  Arms: Mineral water 1
Dietary Supplement: Mineral water (Aso-gun, Kumamoto, Japan)
  Arms: Mineral water 2

SUMMARY:
The purpose of the study is to determine the effect of a specific mineral water on serum lipid concentrations in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as based on medical history and physical examination
* Fasting serum LDL cholesterol > 100 and/or fasting serum triglyceride > 100
* Willing to drink mineral water for 12 weeks
* Willing not to serve as blood donor during the study
* Informed consent signed

Exclusion Criteria:

* Female subjects who are pregnant or nursing a child
* Participation in any clinical trial up to 90 days before Day 01 of this study
* Renal or hepatic dysfunction
* Heart disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-12; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Fasting total cholesterol, LDL cholesterol, and triglyceride levels | Every 4 weeks (Overall 20 weeks)

SECONDARY OUTCOMES:
Fasting serum glucose and HbA1c levels | Every 4 weeks (Overall 20 weeks)
Serum uric acid level | Every 4 weeks (Overall 20 weeks)
Serum adiponectin and leptin levels | Week 0, Week 12
Urinary oxidative stress marker | Week 0, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Fumiko Higashikawa, PhD, Principal Investigator — Hiroshima University
Locations (1):
- Hiroshima University, Hiroshima, Japan